CLINICAL TRIAL: NCT02588911
Title: Randomised Trial of Radiofrequency Ablation vs Conventional Surgery for Superficial Venous Insufficiency: if You Don't Tell, They Won't Know
Brief Title: Radiofrequency Ablation vs Conventional Surgery for Superficial Venous Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nelson Wolosker (Other)
Responsible Party: Sponsor-Investigator, Nelson Wolosker, MD, PhD, Hospital Israelita Albert Einstein
Organization: Hospital Israelita Albert Einstein (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RFA vs CS
Record Dates: First submitted 2015-10-20; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Venous Insufficiency
Keywords: Radiofrequency Catheter Ablation; Operative Surgical Procedure; Saphenous Vein
MeSH Terms: conditions — Venous Insufficiency | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Surgery (Active Comparator): Limb with GSV insufficiency in the same patient, randomised to conventional surgery
  Interventions: Procedure: Conventional Surgery
- Radiofrequency Ablation (Active Comparator): Limb with GSV insufficiency in the same patient, randomised to radiofrequency ablation
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Conventional Surgery — Cranial ligation of the great saphenous vein and branches of the sapheno-femoral junction and stripping of the great saphenous vein
  Arms: Conventional Surgery
Procedure: Radiofrequency Ablation — Catheter-based ablation of the great saphenous vein
  Arms: Radiofrequency Ablation

SUMMARY:
The current study was a double blind randomised controlled trial that compared radiofrequency ablation (RFA) versus conventional surgery (CS) in patients who served as their own controls and who had intact great saphenous veins (GSVs).

DETAILED DESCRIPTION:
Individuals with symptomatic varicose veins and bilateral GSV insufficiency confirmed by duplex ultrasound examination who were candidates for conventional vein stripping were eligible for inclusion in the study. A total of 18 patients entered the trial. As per protocol, each patient was treated with RFA in one leg and CS on the contralateral limb. Randomisation was performed preoperatively using a randomisation table. Patients were not advised of the treatment allocation in order to ensure that this trial was carried out in a blinded fashion. All operations were performed under regional anaesthesia by the same surgical team, skilled in the management of venous disease with extensive expertise in both techniques. Phlebectomy of varicosities was not concomitantly performed.

The independent observer physician not involved in the original operation, the patient, and the duplex ultrasonographer were not aware of the treatment performed in each case and the surgeon was not involved in outcome assessment.

CS. Patients underwent standard procedure of cranial ligation of the GSV and branches of the sapheno-femoral junction (SFJ) using a groin crease incision and stripping of the GSV from SFJ to ankle level, using a vein stripper that was brought out through a small incision near the medial malleolus.

RFA. The procedure was performed under ultrasound guidance. The GSV proximal to the medial malleolus was cannulated with a 7F sheath using surgical cutdown. The tip of the radiofrequency catheter was placed at least 2 cm distal to the SFJ or just distal to the superficial epigastric vein orifice. Patients received tumescent infiltration with cold normal saline (0.9%) circumferentially around the GSV within its enveloping fascia and along the entire length of the treated vein. This was to prevent nerve injury and thermal injury to the skin. Then the catheter was gradually withdrawn according to the device manufacturer's recommendations. The technique consisted of controlled segmental heating of the GSV, using a catheter with a 7-cm heating element (Closure™ system, VNUS Medical Technologies, Inc., San Jose, California, USA). The temperature was maintained at 120° C per segment using a standard time. The thermoablation continued until the catheter tip reached just below the knee. Immediately following treatment with RFA, intraoperative ultrasound imaging was used to confirm shrinkage of the vein.

For limbs operated with the radiofrequency technique, a groin crease incision was made similar to the contralateral side, but with no manipulation of the SFJ. The incision proximal to the medial malleolus was used for sheath insertion. To ensure that the independent observer physician not involved in the original operation, the patient, and the duplex ultrasonographer were not made aware of the treatment done, both incisions were performed on both legs.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Clinical, etiologic, anatomic, pathophysiologic (CEAP): clinical grades 2 to 5 (C2-5), primary (Ep), superficial (As) and reflux only (Pr)
* Duplex scan confirmed primary bilateral GSV insufficiency requiring surgery (insufficiency with reverse venous flow was regarded significant if persisting more than 0.5 seconds in a standing position)
* Duplex scan confirmed suitability for RFA (see exclusion criteria)
* Patients able to give informed consent

Exclusion Criteria:

* Varicose veins without GSV insufficiency on duplex scan
* Previous varicose vein surgery
* Associated small saphenous vein reflux, duplication of the GSV at the SFJ, deep venous insufficiency or previous DVT on duplex scan
* GSV diameter <3 mm or >12 mm in the supine position
* Thrombus in the GSV
* Patients with a pacemaker or internal defibrillator
* Concomitant peripheral arterial disease (ankle-brachial pressure index of <0.9)
* Patients on oral anticoagulants
* Patients with high blood pressure not controlled by medication
* Patients with known thrombophilia, cancer or lupus
* Pregnancy

Ages: 33 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in intensity of hyper pigmentation using a scale of 0 to 10 | One week, one month and six months after surgery
  Patients and physicians were oriented to indicate their subjective perception of intensity of hyperpigmentation on a scale of 0 (no complaint/discomfort) to 10 (maximal complaint/discomfort).
Change in extension of hematoma using a scale of 0 to 10 | One week, one month and six months after surgery
  Patients and physicians were oriented to indicate their subjective perception of extension of hematoma on a scale of 0 (no complaint/discomfort) to 10 (maximal complaint/discomfort).
Change in aesthetic results using a scale of 0 to 10 | One week, one month and six months after surgery
  Patients and physicians were oriented to indicate their subjective perception of aesthetic results on a scale of 0 (unaesthetic) to 10 (excellent results).
Change in pain levels using a scale of 0 to 10 | One week, one month and six months after surgery
  Patients were asked to indicate pain levels on a scale of 0 (no pain) to 10 (worst imaginable pain).
Change in intensity of skin burns using a scale of 0 to 10 | One week, one month and six months after surgery
  Physicians were asked to inform intensity of skin burns on a scale of 0 (no complaint/discomfort) to 10 (maximal complaint/discomfort).
Change in presence of sensitivity alteration | One week, one month and six months after surgery
  Patients were asked to indicate the presence or absence of sensitivity alteration.
Change in presence of thrombophlebitis | One week, one month and six months after surgery
  Physicians were asked to inform the presence or absence of thrombophlebitis.
Change in presence of resection or occlusion of the great saphenous vein | One month, six months and 12 months after surgery
  Duplex ultrasound scan was used to evaluate the presence or absence of resection or occlusion (success rate) of the great saphenous vein.
Change in presence of reflux in the sapheno-femoral junction and in the great saphenous vein | One month, six months and 12 months after surgery
  Duplex ultrasound scan was used to evaluate the presence or absence of reflux in the sapheno-femoral junction and in the great saphenous vein
Change in presence of complications | One month, six months and 12 months after surgery
  Duplex ultrasound scan was used to evaluate the presence or absence of complications such as deep vein thrombosis (DVT) and lymphocele.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Wolosker, MD, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Wittens C, Davies AH, Baekgaard N, Broholm R, Cavezzi A, Chastanet S, de Wolf M, Eggen C, Giannoukas A, Gohel M, Kakkos S, Lawson J, Noppeney T, Onida S, Pittaluga P, Thomis S, Toonder I, Vuylsteke M, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Koncar I, Lindholt J, de Ceniga MV, Vermassen F, Verzini F, Document Reviewers, De Maeseneer MG, Blomgren L, Hartung O, Kalodiki E, Korten E, Lugli M, Naylor R, Nicolini P, Rosales A. Editor's Choice - Management of Chronic Venous Disease: Clinical Practice Guidelines of the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2015 Jun;49(6):678-737. doi: 10.1016/j.ejvs.2015.02.007. Epub 2015 Apr 25. No abstract available. PMID 25920631
- [Background] Siribumrungwong B, Noorit P, Wilasrusmee C, Attia J, Thakkinstian A. A systematic review and meta-analysis of randomised controlled trials comparing endovenous ablation and surgical intervention in patients with varicose vein. Eur J Vasc Endovasc Surg. 2012 Aug;44(2):214-23. doi: 10.1016/j.ejvs.2012.05.017. Epub 2012 Jun 15. PMID 22705163
- [Background] Hinchliffe RJ, Ubhi J, Beech A, Ellison J, Braithwaite BD. A prospective randomised controlled trial of VNUS closure versus surgery for the treatment of recurrent long saphenous varicose veins. Eur J Vasc Endovasc Surg. 2006 Feb;31(2):212-8. doi: 10.1016/j.ejvs.2005.07.005. Epub 2005 Aug 31. PMID 16137898
- [Background] Goode SD, Chowdhury A, Crockett M, Beech A, Simpson R, Richards T, Braithwaite BD. Laser and radiofrequency ablation study (LARA study): a randomised study comparing radiofrequency ablation and endovenous laser ablation (810 nm). Eur J Vasc Endovasc Surg. 2010 Aug;40(2):246-53. doi: 10.1016/j.ejvs.2010.02.026. PMID 20537570
- [Background] Subramonia S, Lees T. Radiofrequency ablation vs conventional surgery for varicose veins - a comparison of treatment costs in a randomised trial. Eur J Vasc Endovasc Surg. 2010 Jan;39(1):104-11. doi: 10.1016/j.ejvs.2009.09.012. Epub 2009 Oct 29. PMID 19879166
- [Derived] Mendes CA, Martins AA, Fukuda JM, Parente JB, Munia MA, Fioranelli A, Teivelis MP, Varella AY, Caffaro RA, Kuzniec S, Wolosker N. Randomized trial of radiofrequency ablation versus conventional surgery for superficial venous insufficiency: if you don't tell, they won't know. Clinics (Sao Paulo). 2016 Nov 1;71(11):650-656. doi: 10.6061/clinics/2016(11)06. PMID 27982166